CLINICAL TRIAL: NCT01389219
Title: Post Partum Maternal and Neonatal Intervention Package: A Cluster Randomized Control Trial in District Sukkur, Pakistan
Brief Title: Post Partum Maternal and Neonatal Intervention Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Pakistan Ministry of Health (Other Government); John Snow, Inc. (Industry); Population Council (Other)
Responsible Party: Dr. Zulfiqar A. Bhutta (Principal investigator), Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 770-Ped/ERC-06
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2007-10

CONDITIONS: Early Postpartum and Newborn Care; Maternal Mortality; Neonatal Mortality
Keywords: Post partum; Neonate; community health care workers
MeSH Terms: conditions — Maternal Death | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control arm
- Intervention clusters (Other): Focus is to increase the number of visits by LHWs to the newborn baby and to ensure that this visit occurs within 48-72 hours of birth. The purpose of this visit was the provision of postpartum maternal and immediate newborn care, including postpartum visit, maternal nutrition supplementation, cord care, eye care, Kangaroo Care, delayed bathing, colostrum administration and linkages to immunization services), complications/illness management through stabilization/referral of cases.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — A comprehensive package of intervention will be developed for the mothers and newborn infants which will be comprised of;
  1. Provision of postpartum maternal and immediate newborn care, including postpartum visit, maternal nutrition supplementation (iron & vitamin A), cord care, eye care, Kangaroo Care, delayed bathing, colostrum administration and linkages to immunization services), complications/illness management through stabilization/referral of cases.
  2. Provision of Information on family planning, birth spacing, LAM counseling, hygiene, danger signs recognition and complications readiness.
  3. Nutrition counseling regarding immediate and exclusive breastfeeding and optimum postpartum diets.
  5. Danger signs of newborn illnesses and maternal complications associated with labor and the postpartum period, care seeking. Early referral for subsequent maternal and newborn morbidities, such as anemia, postpartum depression, fistulas, prolapsed uterus and infections.
  Arms: Intervention clusters

SUMMARY:
Introduction of a community-based intervention package including prevention strategies, early recognition and management of common postpartum & neonatal problems, as well as prompt referral of high risk/complicated cases through trained first level primary health care workers, will result in a significant reduction in Postpartum maternal and neonatal mortality in Pakistan

DETAILED DESCRIPTION:
Introduction of a community-based intervention package including prevention strategies, early recognition and management of common postpartum & neonatal problems, as well as prompt referral of high risk/complicated cases through trained first level primary health care workers, will result in a significant reduction in Postpartum maternal and neonatal mortality in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Neonates delivered within the study area

Exclusion Criteria:

* Neonates delivered outside the study area

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Visit by LHWs | Within 48 - 72 hours of birth
  The aim is to increase the visits of LHWs and examine the newborn within 48- 72 hours of birth

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, MBBS, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Sukkur, Sindh, Pakistan